CLINICAL TRIAL: NCT00946205
Title: Laparoscopic Posterior Rectopexy Without Mesh vs. Laparoscopic Anterior Mesh Rectopexy for Rectal Prolapse - a Prospective, Double-blind, Randomised Study
Brief Title: Laparoscopic Rectopexy for Rectal Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Lene H. Iversen, MD, DMSci, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lap rectopexy 200660096
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Rectal Prolapse
Keywords: rectal prolapse; laparoscopic rectopexy; obstructed defecation
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic anterior mesh rectopexy (Experimental)
  Interventions: Procedure: Laparoscopic anterior mesh rectopexy
- Laparoscopic posterior rectopexy (Active Comparator)
  Interventions: Procedure: Laparoscopic posterior rectopexy

INTERVENTIONS:
Procedure: Laparoscopic posterior rectopexy — The rectum is mobilised down to the os coccygeus, then it is elevated cephalic and sutured with a multifilament suture to the presacral fascia just below the sacral promontory. The lateral stalks should be left intact.
  Arms: Laparoscopic posterior rectopexy
Procedure: Laparoscopic anterior mesh rectopexy — The peritoneum is incised over the right side of the promontory. The incision is extended in an inverted J-form along the right side of rectum and over the deepest part of the pouch of Douglas. Denonvilliers fascia is incised and the rectovaginal (women)/rectovesical (men) septum is broadly opened. A prosthetic mesh (3 x 17 cm) is sutured with nonabsorbable sutures to the ventral aspect of the rectum in the rectovaginal/rectovesical septum and to the lateral seromuscular borders of rectum and fixed upon the promontory using a stapler. The posterior fornix of vagina (women)/floor of the bladder (men) is elevated and sutured to the anterior aspect of the mesh. The incised peritoneum is then closed over the mesh.
  Arms: Laparoscopic anterior mesh rectopexy

SUMMARY:
The aim of the present prospective, double-blind, randomized study is to study whether laparoscopic anterior mesh rectopexy is as good as laparoscopic posterior rectopexy with respect to obstructive defecation afterwards.

DETAILED DESCRIPTION:
Full-thickness rectal prolapse is defined as a "falling down" of the rectum so that it is outside the body. Rectal prolapse can only be treated by surgery.

The choice of procedure depends on the patient's general condition and is based on a clinical judgment. Usually, elderly, high-risk patients are treated by perineal procedures. All other patients are offered an abdominal rectopexy using open or laparoscopic techniques. The general principle for all abdominal procedures is to induce adhesions between the mobilised, elevated rectum and the presacral fascia.

At least 30%-60% develop long-term complications: Obstructive defecation, which may be related to peroperative trauma to rectums innervation. Sparing of the lateral stalks during the rectal mobilisation results in lower frequency of obstructive defecation afterwards, but also higher recurrence rate.

A nerve-sparing laparoscopic technique for rectal prolapse has been developed in Belgium: Laparoscopic anterior mesh rectopexy.

After this procedure, the rate of obstructed defecations afterwards has been reported to less than 10%, that is, much lower than observed after other procedures.

The functional results after this nerve-sparing laparoscopic technique should be compared to those after laparoscopic posterior rectopexy, i.e. the conventional laparoscopic method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with full-thickness rectal prolapse for whom the department otherwise would offer abdominal rectopexy according to the department's recommendation. That is, patient being fit for an abdominal rectopexy procedure.

Exclusion Criteria:

* Age below 18 years.
* Pregnancy or breast-feeding.
* Patients who do not speak or read Danish.
* Dementia or other psychiatric disease, i.e., inability to give informed consent.
* Recurrence of rectal prolapse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-09; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The severity of obstructive defecation as graded by Wexner's incontinence- and constipation-score and Obstructed Defecation Syndrome score | 1 year postoperatively

SECONDARY OUTCOMES:
Physiologic testing of the ano-rectum: Anorectal manometry,anal sensibility,anal ultrasound, colonic transit. | 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Søren Laurberg, Professor, Study Chair — Aarhus University Hospital, Department of Surgery P
Locations (1):
- Aarhus University Hospital, Department of Surgery P, Aarhus, Aarhus C, Denmark

REFERENCES:
- [Background] D'Hoore A, Cadoni R, Penninckx F. Long-term outcome of laparoscopic ventral rectopexy for total rectal prolapse. Br J Surg. 2004 Nov;91(11):1500-5. doi: 10.1002/bjs.4779. PMID 15499644
- [Derived] Lundby L, Iversen LH, Buntzen S, Wara P, Hoyer K, Laurberg S. Bowel function after laparoscopic posterior sutured rectopexy versus ventral mesh rectopexy for rectal prolapse: a double-blind, randomised single-centre study. Lancet Gastroenterol Hepatol. 2016 Dec;1(4):291-297. doi: 10.1016/S2468-1253(16)30085-1. Epub 2016 Oct 4. PMID 28404199